CLINICAL TRIAL: NCT06791603
Title: The Impact of Social Media-delivered Chemotherapy-related Side Effects Education for Breast Cancer Patients Receiving First Time Chemotherapy
Brief Title: The Impact of Social Media-delivered Chemotherapy Side Effects Education for Breast Cancer Patients Receiving Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Pohung Lin, Principal Investigator, clinical pharmacist, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TMU-JIRB N202410024
Record Dates: First submitted 2025-01-11; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Chemotherapy Side Effects; Social Media; Education of Patients
Keywords: pharmacist; chemotherapy education; social media
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized chemotherapy education + video (Experimental): Standardized chemotherapy education+ video
  Interventions: Other: Standardized chemotherapy education + video
- Chemotherapy handouts (No Intervention): Chemotherapy handouts

INTERVENTIONS:
Other: Standardized chemotherapy education + video — Videos will be provided with patients and they will watch videos during the visit. The information regarding the prevention and management of side effects and further instructions when to visit hospital. Patients will have access to videos and watch videos after leaving the hospital for the entire treatment course
  Arms: Standardized chemotherapy education + video

SUMMARY:
The goal of this clinical trial is to learn if a standardized pharmacists-provided education module by social media can improve patients' knowledge of chemotherapy-related side effects. The main questions it aims to answer is:

• Do patients who received a standardized pharmacists-provided education module by social media improve their knowledge of chemotherapy-related side effects? Researchers will compare standardized chemotherapy education +video (experimental group) versus chemotherapy handouts (control group).

Participants will:

* Received standardized chemotherapy education + video or chemotherapy handouts at the first and second chemotherapy section.
* Fill out a questionnaire for outcomes assessment.

DETAILED DESCRIPTION:
The pharmacist-provided video education model for patients undergoing first time chemotherapy was developed. The content of the education video included the mechanism of side effects, its recognition, preventive measures, non-medical management, and further instructions when to visit hospital were included.

Patients were randomly assigned into two groups with different education strategies:

Standardized chemotherapy education +video (experimental group) versus chemotherapy handouts (control group). Every patient was asked to fill out a questionnaire prior to the implementation of the education model in both groups. The pre-test questionnaires consisted of baseline knowledge and personal information. Patients in the experimental group would receive standardized chemotherapy education by pharmacists, including chemotherapy regimen, the purpose of chemotherapy, the number of cycles, duration of chemotherapy and the common side effects of chemotherapy on the first day of chemotherapy cycle. Videos will be provided with patients and they will watch videos during the visit. The information regarding the prevention and management of side effects and further instructions when to visit hospital. Patients will have access to videos and watch videos after leaving the hospital for the entire treatment course. The education time will be last around 15 to 20 minutes. In terms of control group, pharmacists will briefly explain and provide chemotherapy handouts, including chemotherapy regimen, the purpose of chemotherapy, the number of cycles, duration of chemotherapy and the common side effects of chemotherapy. The duration of visit will be around 5 to 10 minutes. After the education section, patients will be asked to do a post-test questionnaire of their knowledge and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients aged 18 or older undergoing their first chemotherapy.
* Possess a smartphone and are able to watch videos on it.

Exclusion Criteria:

* Unable to read or complete questionnaires in Chinese.
* Cognitive impairments.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
A questionnaire with 5 questions of side effects management | 1. First time receiving chemotherapy 2. Second time receiving chemotherapy (3 to 4 weeks depend on schedule)
  Each question is a multiple choice with 4 options and 1 correct answer

SECONDARY OUTCOMES:
FACT-B, The Functional Assessment of Cancer Therapy - Breast | 1. First time receiving chemotherapy 2. Second time receiving chemotherapy (3 to 4 weeks depend on schedule)

CONTACTS AND LOCATIONS:
Overall Officials: Pohung Lin, PharmD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No